CLINICAL TRIAL: NCT03014492
Title: Novel Protection Against Potential Brain Injury During Competitive Non-helmeted Sport in Females
Brief Title: Concussion Prevention in Female Soccer Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2016-0988
Record Dates: First submitted 2017-01-05; First posted 2017-01-09 (Estimated); Results first posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-09

CONDITIONS: Concussion, Mild; Concussion, Brain
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collar Group (Experimental): Soccer girls that wore the collar device
  Interventions: Device: Q Collar
- No Collar Group (No Intervention): soccer girls that did not wear the collar

INTERVENTIONS:
Device: Q Collar — Collar designed to mitigate slosh in the brain
  Arms: Collar Group

SUMMARY:
The purpose of the study is to monitor longitudinal changes in brain structure and function between the preseason and postseason, in a population of soccer playing athletes wearing the Device and compared to a similar population not wearing the device. Secondly, the purpose is to determine the protection of the device relative to amount and magnitude of sustained head impacts.

DETAILED DESCRIPTION:
This study will investigate the effectiveness of this device in high school athletes playing a non-helmeted sport such as soccer. Athletes participating in this study will be randomly assigned to one of two groups: 1) Device wearing during the season or 2) Non-device wearing during the season. This study will focus on the use and effectiveness of the device solely in females, as male football and hockey players have previously been investigated. All participants will be outfitted with an adhesive patch-like accelerometer (which will be placed behind the ear (Xpatch-X2 Biosystems http://www.x2biosystems.com/x2_x_patch/) which will measure the magnitude of every impact to the head sustained by the athlete. Effectiveness of the device will be determined via differences in longitudinal brain imaging and functional testing following competitive soccer participation. A subset of athletes who report a diagnosed concussion will also receive additional brain neuroanatomical and neurophysiological testing within a week following the diagnosed concussive event. At each of these time points participants will also undergo various neurocognitive assessments

ELIGIBILITY:
Inclusion Criteria:

* Female
* Normal healthy volunteer
* Able to provide written consent
* Must be 14 years or older and a participant on a high school soccer team

Exclusion Criteria:

* Unable to provide written consent
* History of neurological deficits, previous cerebral infarction, or severe head trauma as indicated through pre-season screening:
* Medical contraindications to restriction of venous outflow via the internal jugular veins (known increased intracerebral pressure, metabolic acidosis or alkalosis)
* Glaucoma (Narrow Angle or Normal Tension)
* Hydrocephalus
* Recent penetrating brain trauma (within 6 months)
* Known carotid hypersensitivity
* Known increased intracranial pressure
* Central vein thrombosis
* Any known airway obstruction
* Any known seizure disorder

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Myer, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinanti Childrens Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Collar Group | No Collar Group
Started | 44 | 28
Completed | 44 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Collar Group | No Collar Group | Total
Number analyzed (Participants) | 44 | 28 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44 | 28 | 72
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 28 | 72
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 44 | 28 | 72
Age of participant [Mean (Standard Deviation); unit: years] | 16.06 (1.10) | 15.95 (1.04) | 16.0 (1.07)

OUTCOME MEASURES:

1. Primary Outcome: Pre-season to Post-season DTI Percentage Change
Description: Determine % changes in brain structure between pre-season and post-season in AD, axial diffusivity; FA, fractional anisotropy; MD, mean diffusivity; RD, radial diffusivity.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Collar Group | No Collar Group
Number analyzed (Participants) | 24 | 22
percentage of change
  FA | -0.17 (1.99) | -1.27 (1.35)
  MD | 0.45 (2.23) | 2.83 (2.46)
  AD | 0.37 (2.23) | 2.58 (2.34)
  RD | 0.53 (2.72) | 3.52 (2.6)

2. Primary Outcome: Number of Participants Completing EEG
Description: Number of participants completing EEG
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Collar Group | No Collar Group
Number analyzed (Participants) | 44 | 28
Participants | 44 | 28

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Collar Group | No Collar Group
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/28
Other Adverse Events (participants affected / at risk) | 0/44 | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT03014492/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-03-01): https://cdn.clinicaltrials.gov/large-docs/92/NCT03014492/Prot_SAP_001.pdf